CLINICAL TRIAL: NCT06117436
Title: Impact of Cilostazol Versus Cilostazol and Selenium Combination on the Healing of Diabetic Foot Ulcer Patients: a Randomized Controlled Trial
Brief Title: Impact of Cilostazol Versus Cilostazol and Selenium Combination on the Healing of Diabetic Foot Ulcer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hadeer Eid Eliwa Ibrahim Fadel, Assistant Lecturer, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSDFU81
Record Dates: First submitted 2023-10-19; First posted 2023-11-07 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Wound Heal
MeSH Terms: interventions — Cilostazol; Selenium

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): patients will receive standard wound care and diabetes management (that includes bed rest with elevation, antibiotics, analgesics, and dressings).
- Cilostazol Group (Active Comparator): patients will receive Cilostazol 100 mg tablets per oral once daily in addition to standard wound care and diabetes management.
  Interventions: Drug: Cilostazol
- Cilostazol & Selenium Group (Active Comparator): Cilostazol 100 mg tablets plus Selenium 200 mcg tablets per oral once daily, in addition to standard wound care and diabetes management.
  Interventions: Drug: Cilostazol; Drug: Selenium

INTERVENTIONS:
Drug: Cilostazol — Cilostazol 100 MG oral tablet once daily antiplatelet, Selenium 200mcg tablet once daily, anti oxidant
  Other Names: cilosort
  Arms: Cilostazol & Selenium Group; Cilostazol Group
Drug: Selenium — Selenium 200 mcg oral tablet once daily
  Arms: Cilostazol & Selenium Group

SUMMARY:
The growing incidence of DM can lead to the increased prevalence of diabetic foot complications, which have become a serious medical, social, and economic concern of global importance. this study aims to find a novel intervention that improve wound healing in diabetic foot ulcer to improve patients' quality of life, reduce amputation rate, and reduce the mortality rate among diabetic foot ulcer patients

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be adult diabetic patients aged 18 years and older with non-ischemic diabetic foot ulcers Wagner's grade 2, 3, and 4.

Exclusion Criteria:

1. Wagner's grade 5 patients (because of the indications for amputation).
2. Patients with poor glycemic control at the time of inclusion (HbA1c>12%).
3. Patients who need either direct graft or indirect revascularization procedure during the study.
4. Patients with Cilostazol or Selenium allergy.
5. Patients with Cilostazol contraindications (Heart Failure, bleeding disorder).
6. Patients with a history of comorbidities that interfere with wound healing (cancers, congestive heart failure, end-stage renal disease, and liver failure).
7. Presence of clinical signs of active infection unresponsive to oral antibiotics (oedema, erythema, discharge, regional lymph node enlargement, pain, or fever).
8. Patients who take medications that interfere with wound healing (glucocorticoids, immunosuppressive and cytotoxic drugs) at the time of inclusion.
9. Non-diabetic patients with foot wounds due to vascular or dermatological reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Wound Healing size | 3 months
  ulcer length, width, and depth in Cm

SECONDARY OUTCOMES:
Effect on Matrix Metalloproteinase-9 (MMP-9) level | 3 months
  will be used by ELISA Kit
Occurrence of infection | 3 months
  any symptoms of infection Include (Redness, Edema and pain at the site of infection)
Treatment-related side effects. | 3 months
  by asking the patient by phone call

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Diabetes and Endocrinology, Cairo, Egypt

REFERENCES:
- [Derived] Eliwa HE, Wakeel LME, Mahfouz AA, Sayed R. Impact of Cilostazol versus Cilostazol and Selenium Combination on The Healing of Diabetic Foot Ulcer Patients: A Randomized Controlled Trial. Diabetol Metab Syndr. 2026 Jan 6;18(1):36. doi: 10.1186/s13098-025-02053-4. PMID 41495844